CLINICAL TRIAL: NCT06009289
Title: Application of Precision Medicine to Phototherapy: a Stepped Care Approach to Consolidate Sleep and Slow Cognitive Decline in Older Adults
Brief Title: Light and Sleep Fragmentation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Professor, Stanford University
Organization: VA Palo Alto Health Care System (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-71788
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Sleep; Mild Cognitive Impairment; Mood Disorders
MeSH Terms: conditions — Cognitive Dysfunction; Mood Disorders | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): One hour of daily bright light exposure beginning one hour after wake time.
  Interventions: Behavioral: Light therapy
- Stepped care (Experimental): One hour of daily bright light exposure in the afternoon
  Interventions: Behavioral: Light therapy

INTERVENTIONS:
Behavioral: Light therapy — One hour of exposure to bright light, either by being outdoors or with a phototherapy lamp if indoor

SUMMARY:
This trial will examine scheduled exposure to bright light in the morning and afternoon as a countermeasure to sleep fragmentation in older individuals with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment
* Age >65

Exclusion Criteria:

* Severe depression
* Unstable psychiatric or medical disease
* Acute infection

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Sleep fragmentation | 4 weeks
  24 hour sleep wake patterns will be quantitated with a non-parametric measure, intradaily variation

SECONDARY OUTCOMES:
Cognition | 6 months
  Performance on the WAIS-4
Mood | 6 months
  Geriatric Depression Scale, range: 0-15 with higher scores being associated with greater depressive symptomatology

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of study and publication of data, deidentified IPD will be uploaded to Dryad with documentation. Analytic code will be shared with Github
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: within six months after publication; no restrictions on duration of availability
URL: https://laneguides.stanford.edu/DataManagement/Sharing